CLINICAL TRIAL: NCT02915016
Title: A Phase 1/2a Clinical Trial to Evaluate the Safety and Immunogenicity of HIV Clade C DNA, and of MF59®- or AS01B-Adjuvanted Clade C Env Protein in Various Combinations, in Healthy, HIV-Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of HIV Clade C DNA Vaccine and MF59- or AS01B-Adjuvanted Clade C Env Protein Vaccines in Various Combinations in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 108; 12007 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 (Experimental): Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo in their right deltoid at Months 0 and 1, and placebo and the Protein/MF59 vaccine in their right deltoid at Months 3 and 6.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Bivalent Subtype C gp120/MF59 vaccine; Biological: Placebo
- Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B (Experimental): Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo in their right deltoid at Months 0 and 1, and placebo and the Protein/AS01B vaccine in their right deltoid at Months 3 and 6.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Bivalent Subtype C gp120/AS01B vaccine; Biological: Placebo
- Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B (Experimental): Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo in their right deltoid at Months 0 and 1, and placebo and the Protein/AS01B vaccine in their right deltoid at Months 3 and 6.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Bivalent Subtype C gp120/AS01B vaccine; Biological: Placebo
- Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 (Experimental): Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, and 6 and placebo in their left deltoid at Month 3. They will receive placebo and the Protein/MF59 vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Bivalent Subtype C gp120/MF59 vaccine; Biological: Placebo
- Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B (Experimental): Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, and 6 and placebo in their left deltoid at Month 3. They will receive placebo and the Protein/AS01B vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Bivalent Subtype C gp120/AS01B vaccine; Biological: Placebo
- Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B (Experimental): Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, and 6 and placebo in their left deltoid at Month 3. They will receive placebo and the Protein/AS01B vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: Bivalent Subtype C gp120/AS01B vaccine; Biological: Placebo
- Group 7: Placebo + Protein/AS01B (Experimental): Participants will receive placebo in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo and the Protein/AS01B vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3.
  Interventions: Biological: Bivalent Subtype C gp120/AS01B vaccine; Biological: Placebo
- Group 8: Placebo (Placebo Comparator): Participants will receive placebo in both their right and left deltoids at Months 0, 1, 3, and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DNA-HIV-PT123 vaccine — Contains a mixture of three DNA plasmids in a 1:1:1 ratio, each at 1.33 mg: 1) clade C 96ZM651 gag, 2) clade C 96ZM651 gp140, and 3) clade C CN54 pol-nef, delivered at a total dose of 4 mg, administered by intramuscular (IM) injection to the left deltoid as a single 1 mL dose.
  Arms: Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59; Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59; Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B
Biological: Bivalent Subtype C gp120/MF59 vaccine — Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, each at a dose of 100 mcg, mixed with MF59 adjuvant, administered by IM injection to the right deltoid as a single 0.5 mL dose.
  Other Names: Protein/MF59 vaccine
  Arms: Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59; Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59
Biological: Bivalent Subtype C gp120/AS01B vaccine — Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, mixed with AS01B adjuvant, administered by IM injection to the right deltoid as a single 0.75 mL dose.
  Groups 2 and 5 will receive a 100 mcg dose. Groups 3, 6, and 7 will receive a 20 mcg dose.
  Other Names: Protein/AS01B vaccine
  Arms: Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 7: Placebo + Protein/AS01B
Biological: Placebo — Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.

SUMMARY:
This study will evaluate the safety and immune response to the DNA-HIV-PT123 vaccine used in combination with one of two protein vaccines (Bivalent Subtype C gp120/MF59 or Bivalent Subtype C gp120/AS01B) in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and immune response of the DNA-HIV-PT123 vaccine when used in combination with one of two protein vaccines: Bivalent Subtype C gp120/MF59 (Protein/MF59) or Bivalent Subtype C gp120/AS01B (Protein/AS01B). These protein vaccines may boost the immune response to the DNA vaccine.

The study will enroll healthy, HIV-uninfected adults. Participants will be randomly assigned to one of eight groups, and each group will receive a different sequence of vaccines during the study. Groups 1 and 4 will receive the DNA-HIV-PT123 vaccine, the Protein/MF59 vaccine, and placebo. Groups 2, 3, 5, 6, and 7 will receive the DNA-HIV-PT123 vaccine, the Protein/AS01B vaccine, and placebo. Group 8 will only receive placebo.

All participants will receive their assigned vaccines at Months 0, 1, 3, and 6. Each of these visits will include three injections. Follow-up visits will occur at Week 2 and Months 1.5, 3.5, 6.25, 6.5, 9, and 12.

Study visits will include a physical examination, an interview and/or questionnaire, HIV testing and HIV risk reduction counseling, and urine and blood collection. Participants may optionally choose to provide stool, rectal fluid, cervical fluid, or semen samples. Participants will be contacted 6 months after the last scheduled visit by phone, text message, or e-mail for information about their health.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 40 years
* Access to a participating HVTN clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit
* Willing to be contacted by phone, text message, or e-mail 6 months after completion of the scheduled clinic visits
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

Laboratory Inclusion Values:

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: ALT, AST, and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA). Non-US sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.

Reproductive status:

United States

A volunteer who was born female must:

* Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in the United States is defined as using any 1 or more of the following methods:

  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy), or
  * Any other contraceptive method approved by the HVTN 108 protocol safety review team (PSRT)
* Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
* Or be sexually abstinent.

Southern Africa

A volunteer who was born female must:

* Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in Southern Africa is defined as using 2 methods of birth control. These include 1 of the following methods:

  * Condoms (male or female)
  * Diaphragm or cervical cap
* PLUS 1 of the following methods:

  * IUD,
  * Hormonal contraception (in accordance with applicable national contraception guidelines), or
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy), or
  * Any other contraceptive method approved by the HVTN 108 PSRT
* Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
* Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Other

Volunteers 21 years of age and older who were born female consenting to provide cervical samples:

* Pap smear within:

  * the 3 years prior to enrollment with the latest result reported as normal or atypical squamous cells of undetermined significance (ASCUS), or
  * the 5 years prior to enrollment, with the latest result reported as normal, or ASCUS with no evidence of high risk human papillomavirus (HPV).
* If no pap smear was done within the last 3 years (or within the last 5 years, if high risk HPV testing was performed), the volunteer must be willing to undergo a pap smear with the result reported as normal or ASCUS prior to sample collection.

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 108 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and Other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 108 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 108 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 108 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency

Clinically significant medical conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent US National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Garrett, Study Chair — Centre for the AIDS Programme of Research in South Africa
Locations (17):
- United States (8):
  - Alabama CRS, Birmingham, Alabama
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- South Africa (9):
  - Kliptown Soweto CRS, Johannesburg, Gauteng
  - The Aurum Institute Tembisa Clinical Research Centre CRS, Johannesburg, Gauteng
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - Setshaba Research Centre CRS, Soshanguve, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic CRS, Ladysmith, KwaZulu-Natal
  - Verulam CRS, Verulam, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
  - Emavundleni CRS, Cape Town, Western Cape

REFERENCES:
- [Derived] Conley HE, Oh SY, Garrett N, Kublin J, Monaco CL, Watts S, Jha S, Ferrari G, Tomaras GD, Geraghty DE, Chan C, Pollara J. IgG and Fc Receptor Genetic Variation Associates With Functional Antibody Responses in a DNA and Protein Candidate HIV Vaccine Trial. J Acquir Immune Defic Syndr. 2025 Dec 1;100(4):371-375. doi: 10.1097/QAI.0000000000003734. PMID 40704585
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Garrett N, Dintwe O, Monaco CL, Jones M, Seaton KE, Church EC, Grunenberg N, Hutter J, deCamp A, Huang Y, Lu H, Mann P, Robinson ST, Heptinstall J, Jensen RL, Pantaleo G, Ding S, Koutsoukos M, Hosseinipour MC, Van Der Meeren O, Gilbert PB, Ferrari G, Andersen-Nissen E, McElrath MJ, Tomaras GD, Gray GE, Corey L, Kublin JG; HVTN 108 and HVTN 111 Study Teams. Safety and Immunogenicity of a DNA Vaccine With Subtype C gp120 Protein Adjuvanted With MF59 or AS01B: A Phase 1/2a HIV-1 Vaccine Trial. J Acquir Immune Defic Syndr. 2024 Aug 1;96(4):350-360. doi: 10.1097/QAI.0000000000003438. Epub 2024 Jun 21. PMID 38916429
- [Derived] Hanass-Hancock J, Carpenter B, Reddy T, Nzuza A, Gaffoor Z, Goga A, Andrasik M. Participants' characteristics and motivations to screen for HIV vaccine and monoclonal antibody trials in KwaZulu-Natal, South Africa. Trials. 2021 Dec 11;22(1):897. doi: 10.1186/s13063-021-05792-7. PMID 34895272
- [Derived] Mngadi KT, Maharaj B, Duki Y, Grove D, Andriesen J. Using Mobile Technology (pMOTAR) to Assess Reactogenicity: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 3;7(10):e175. doi: 10.2196/resprot.9396. PMID 30282622

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B: Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo in their right deltoid at Months 0 and 1, and placebo and the Protein/AS01B vaccine in their right deltoid at Months 3 and 6.
  DNA-HIV-PT123 vaccine: Contains a mixture of three DNA plasmids in a 1:1:1 ratio, each at 1.33 mg: 1) clade C 96ZM651 gag, 2) clade C 96ZM651 gp140, and 3) clade C CN54 pol-nef, delivered at a total dose of 4 mg, administered by intramuscular (IM) injection to the left deltoid as a single 1 mL dose.
  Bivalent Subtype C gp120/AS01B vaccine: Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, mixed with AS01B adjuvant, administered by IM injection to the right deltoid as a single 0.75 mL dose.
  Groups 2 and 5 will receive a 100 mcg dose. Groups 3, 6, and 7 will receive a 20 mcg dose.
  Placebo: Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.
- Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B; Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B: Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, and 6 and placebo in their left deltoid at Month 3. They will receive placebo and the Protein/AS01B vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3.
  DNA-HIV-PT123 vaccine: Contains a mixture of three DNA plasmids in a 1:1:1 ratio, each at 1.33 mg: 1) clade C 96ZM651 gag, 2) clade C 96ZM651 gp140, and 3) clade C CN54 pol-nef, delivered at a total dose of 4 mg, administered by intramuscular (IM) injection to the left deltoid as a single 1 mL dose.
  Bivalent Subtype C gp120/AS01B vaccine: Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, mixed with AS01B adjuvant, administered by IM injection to the right deltoid as a single 0.75 mL dose.
  Groups 2 and 5 will receive a 100 mcg dose. Groups 3, 6, and 7 will receive a 20 mcg dose.
  Placebo: Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.
- Group 7: Placebo + Protein/AS01B: Participants will receive placebo in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo and the Protein/AS01B vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3.
  Bivalent Subtype C gp120/AS01B vaccine: Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, mixed with AS01B adjuvant, administered by IM injection to the right deltoid as a single 0.75 mL dose.
  Groups 2 and 5 will receive a 100 mcg dose. Groups 3, 6, and 7 will receive a 20 mcg dose.
  Placebo: Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.
Period: Overall Study
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Started | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Month 6.5 Immunogenicity Timepoint (HIV uninfected at Month 6.5 and specimen available for assays) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
Completed | 23 | 47 | 42 | 26 | 43 | 44 | 38 | 20
Not Completed | 7 | 3 | 8 | 4 | 7 | 6 | 12 | 4
Not completed — Lost to Follow-up | 4 | 2 | 5 | 3 | 5 | 2 | 8 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 1 | 3 | 1 | 1
Not completed — Elected not to continue | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — HIV infection | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Participant unable to adhere | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59: Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, 3, and 6. They will receive placebo in their right deltoid at Months 0 and 1, and placebo and the Protein/MF59 vaccine in their right deltoid at Months 3 and 6. DNA-HIV-PT123 vaccine: Contains a mixture of three DNA plasmids in a 1:1:1 ratio, each at 1.33 mg: 1) clade C 96ZM651 gag, 2) clade C 96ZM651 gp140, and 3) clade C CN54 pol-nef, delivered at a total dose of 4 mg, administered by intramuscular (IM) injection to the left deltoid as a single 1 mL dose. Bivalent Subtype C gp120/MF59 vaccine: Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, each at a dose of 100 mcg, mixed with MF59 adjuvant, administered by IM injection to the right deltoid as a single 0.5 mL dose. Placebo: Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.
- Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59: Participants will receive the DNA-HIV-PT123 vaccine in their left deltoid at Months 0, 1, and 6 and placebo in their left deltoid at Month 3. They will receive placebo and the Protein/MF59 vaccine in their right deltoid at Months 0, 1, and 6 and placebo in their right deltoid at Month 3. DNA-HIV-PT123 vaccine: Contains a mixture of three DNA plasmids in a 1:1:1 ratio, each at 1.33 mg: 1) clade C 96ZM651 gag, 2) clade C 96ZM651 gp140, and 3) clade C CN54 pol-nef, delivered at a total dose of 4 mg, administered by intramuscular (IM) injection to the left deltoid as a single 1 mL dose. Bivalent Subtype C gp120/MF59 vaccine: Clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, each at a dose of 100 mcg, mixed with MF59 adjuvant, administered by IM injection to the right deltoid as a single 0.5 mL dose. Placebo: Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.
- Group 8: Placebo: Participants will receive placebo in both their right and left deltoids at Months 0, 1, 3, and 6. Placebo: Sodium Chloride, 0.9%, administered by IM injection at volumes to match the active products.
- Total: Total of all reporting groups
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo | Total
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24 | 334
Age, Continuous [Median (Full Range); unit: years] | 24 [18 to 40] | 25 [18 to 39] | 25 [18 to 40] | 24 [18 to 38] | 27 [18 to 39] | 25 [18 to 38] | 25 [18 to 39] | 26 [19 to 39] | 25 [18 to 40]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 6 | 9 | 5 | 4 | 6 | 9 | 7 | 3 | 49
  21 - 30 years | 20 | 35 | 39 | 22 | 32 | 33 | 36 | 16 | 233
  31 - 40 years | 4 | 6 | 6 | 4 | 12 | 8 | 7 | 5 | 52
  41 - 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Over 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 19 | 22 | 24 | 18 | 30 | 25 | 22 | 13 | 173
    Male | 11 | 28 | 26 | 12 | 20 | 25 | 28 | 11 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 4 | 1 | 3 | 6 | 3 | 0 | 26
  Not Hispanic or Latino | 24 | 47 | 46 | 29 | 47 | 44 | 47 | 24 | 308
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 5
  Asian | 4 | 3 | 3 | 4 | 5 | 4 | 2 | 0 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 27 | 29 | 9 | 26 | 24 | 27 | 11 | 161
  White | 18 | 19 | 16 | 17 | 18 | 17 | 16 | 13 | 134
  More than one race | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 27 | 27 | 26 | 27 | 27 | 27 | 15 | 202
  Africa | 4 | 23 | 23 | 4 | 23 | 23 | 23 | 9 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 7 days after each vaccine dose at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Pain: None | 5 | 7 | 6 | 8 | 10 | 5 | 4 | 10
  Pain: Mild | 21 | 20 | 27 | 19 | 24 | 18 | 24 | 13
  Pain: Moderate | 4 | 23 | 17 | 3 | 16 | 27 | 22 | 1
  Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain: Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tenderness: None | 4 | 8 | 11 | 5 | 8 | 9 | 6 | 8
  Tenderness: Mild | 20 | 16 | 16 | 21 | 23 | 20 | 17 | 16
  Tenderness: Moderate | 6 | 26 | 23 | 4 | 18 | 21 | 27 | 0
  Tenderness: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Tenderness: Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 2 | 6 | 5 | 4 | 8 | 4 | 4 | 7
  Pain and/or Tenderness: Mild | 21 | 16 | 22 | 22 | 21 | 16 | 18 | 16
  Pain and/or Tenderness: Moderate | 7 | 28 | 23 | 4 | 20 | 30 | 28 | 1
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Pain and/or Tenderness: Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 7 days after each vaccine dose at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Erythema: None | 26 | 35 | 38 | 23 | 34 | 36 | 31 | 21
  Erythema: Not gradable | 3 | 4 | 4 | 3 | 3 | 4 | 5 | 2
  Erythema: Grade 1: Less than 5 cm diameter | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
  Erythema: Grade 1: Between 6.25 to 25 cm sq area | 1 | 2 | 2 | 0 | 3 | 2 | 3 | 0
  Erythema: Grade 2: Between 5 to 10 cm diameter | 0 | 1 | 0 | 1 | 3 | 0 | 2 | 1
  Erythema: Grade 2: Between 25 to 100 cm sq area | 0 | 4 | 2 | 3 | 5 | 3 | 6 | 0
  Erythema: Grade 3: Greater or equal to 10 cm | 0 | 2 | 1 | 0 | 1 | 3 | 2 | 0
  Erythema: Grade 3: Greater or equal to 100 cm sq | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
  Erythema: Grade 3: complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: Grade 4: complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration: None | 28 | 35 | 37 | 23 | 33 | 38 | 36 | 24
  Induration: Not gradable | 1 | 6 | 7 | 2 | 4 | 2 | 4 | 0
  Induration: Grade 1: Less than 5 cm diameter | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
  Induration: Grade 1: Between 6.25 to 25 cm sq area | 0 | 2 | 2 | 2 | 5 | 3 | 6 | 0
  Induration: Grade 2: Between 5 to 10 cm diameter | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Induration: Grade 2: Between 25 to 100 cm sq area | 1 | 5 | 3 | 2 | 4 | 3 | 2 | 0
  Induration: Grade 3: Greater or equal to 10 cm | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0
  Induration: Grade 3: Greater or equal to 100 cm sq | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Induration: Grade 3: complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration: Grade 4: complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 25 | 31 | 34 | 22 | 31 | 35 | 30 | 21
  Erythema and/or Induration: Not gradable | 3 | 7 | 7 | 2 | 4 | 4 | 4 | 2
  Erythema and/or Induration: Grade 1: Less than 5 cm diameter | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
  Erythema and/or Induration: Grade 1: Between 6.25 to 25 cm sq area | 1 | 3 | 3 | 2 | 4 | 3 | 5 | 0
  Erythema and/or Induration: Grade 2: Between 5 to 10 cm diameter | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 1
  Erythema and/or Induration: Grade 2: Between 25 to 100 cm sq area | 1 | 4 | 2 | 3 | 6 | 3 | 6 | 0
  Erythema and/or Induration: Grade 3: Greater or equal to 10 cm | 0 | 2 | 1 | 0 | 1 | 3 | 2 | 0
  Erythema and/or Induration: Grade 3: Greater or equal to 100 cm sq | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
  Erythema and/or Induration: Grade 3: complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Grade 4: complications | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Reaction is the maximum of the individual systemic variables for a participant. It does not include temperature.
Time Frame: Measured through 7 days after each vaccination at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Malaise and/or fatigue: None | 14 | 20 | 18 | 18 | 16 | 11 | 16 | 15
  Malaise and/or fatigue: Mild | 11 | 21 | 15 | 10 | 18 | 14 | 10 | 5
  Malaise and/or fatigue: Moderate | 4 | 8 | 14 | 1 | 13 | 21 | 23 | 4
  Malaise and/or fatigue: Severe | 1 | 1 | 3 | 1 | 3 | 4 | 1 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 17 | 24 | 20 | 16 | 23 | 15 | 17 | 18
  Myalgia: Mild | 9 | 16 | 15 | 11 | 11 | 11 | 12 | 4
  Myalgia: Moderate | 4 | 10 | 15 | 3 | 14 | 22 | 20 | 2
  Myalgia: Severe | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 20 | 21 | 15 | 14 | 18 | 14 | 13 | 13
  Headache: Mild | 7 | 21 | 21 | 11 | 18 | 14 | 17 | 8
  Headache: Moderate | 3 | 7 | 14 | 4 | 11 | 21 | 20 | 2
  Headache: Severe | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 1
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 21 | 37 | 34 | 22 | 38 | 30 | 30 | 20
  Nausea: Mild | 7 | 12 | 11 | 6 | 8 | 13 | 10 | 3
  Nausea: Moderate | 2 | 1 | 5 | 2 | 4 | 7 | 10 | 1
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting: None | 29 | 46 | 47 | 29 | 45 | 45 | 42 | 20
  Vomiting: Mild | 1 | 3 | 2 | 1 | 5 | 5 | 4 | 3
  Vomiting: Moderate | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1
  Vomiting: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 27 | 34 | 32 | 25 | 25 | 22 | 23 | 21
  Chills: Mild | 3 | 9 | 8 | 5 | 12 | 8 | 6 | 3
  Chills: Moderate | 0 | 6 | 9 | 0 | 11 | 19 | 17 | 0
  Chills: Severe | 0 | 1 | 1 | 0 | 2 | 1 | 4 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 25 | 38 | 33 | 26 | 29 | 26 | 24 | 20
  Arthralgia: Mild | 5 | 9 | 12 | 4 | 15 | 10 | 10 | 4
  Arthralgia: Moderate | 0 | 3 | 5 | 0 | 5 | 12 | 15 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 12 | 13 | 8 | 8 | 11 | 3 | 8 | 9
  Max. Systemic Symptoms: Mild | 10 | 19 | 19 | 13 | 16 | 12 | 15 | 10
  Max. Systemic Symptoms: Moderate | 7 | 17 | 19 | 7 | 19 | 31 | 22 | 4
  Max. Systemic Symptoms: Severe | 1 | 1 | 4 | 2 | 4 | 4 | 5 | 1
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 29 | 41 | 38 | 26 | 37 | 39 | 36 | 22
  Temperature: Mild | 1 | 4 | 9 | 2 | 8 | 6 | 6 | 2
  Temperature: Moderate | 0 | 5 | 2 | 1 | 3 | 4 | 6 | 0
  Temperature: Severe | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0

4. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: For participants reporting multiple AEs over the time frame, the maximum relationship is counted.
Time Frame: Measured through 30 days after each vaccination at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Related | 3 | 2 | 1 | 5 | 4 | 4 | 2 | 1
  Not Related | 21 | 32 | 33 | 15 | 35 | 27 | 25 | 12
  No AE reported | 6 | 16 | 16 | 10 | 11 | 19 | 23 | 11

5. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: For participants reporting multiple AEs over the time frame, the maximum severity grade is counted.
Time Frame: Measured through 30 days after each vaccination at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Mild | 11 | 13 | 10 | 6 | 19 | 8 | 9 | 3
  Moderate | 12 | 19 | 22 | 10 | 16 | 22 | 16 | 10
  Severe | 1 | 2 | 2 | 4 | 3 | 1 | 2 | 0
  Potentially life-threatening | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  No AE reported | 6 | 16 | 16 | 10 | 11 | 19 | 23 | 11

6. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Measured as outlined in Version 2.0 (January 2010) of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual)
Time Frame: Measured through Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0

7. Primary Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs)
Description: There were no adverse events of special interest reported by any participant.
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants Reporting New Chronic Conditions (Requiring Medical Intervention for ≥ 30 Days)
Description: There were no new chronic conditions (requiring medical intervention for ≥ 30 days) reported by any participant.
Time Frame: Measured through Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: There were no early study terminations associated with an AE or reactogenicity reported by any participant.
Time Frame: Measured through Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm.
Time Frame: Measured through Month 6.5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Clinical event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reactogenicity symptom | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 0
  Other reason | 3 | 2 | 2 | 1 | 1 | 4 | 1 | 3
  No Discontinuation | 26 | 48 | 48 | 28 | 47 | 43 | 43 | 21

11. Primary Outcome: Chemistry and Hematology Laboratory Measures - ALT(SGPT), AST, Alkaline Phosphatase.
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 1, 3, and 6
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
U/L
  ALT (SGPT) (U/L)-Screening | 15 [12 to 18] | 14.5 [12 to 20] | 15 [11 to 18] | 13.5 [11 to 20] | 16.5 [13 to 25] | 16 [11 to 23] | 15 [12 to 21] | 17 [12 to 20]
  ALT (SGPT) (U/L)-Day 14 | 14 [12.5 to 16.5] | 16 [11 to 19] | 16 [12 to 21] | 13 [10 to 19] | 17.5 [13 to 24] | 16 [11 to 23.5] | 15.5 [10 to 19.5] | 16 [11 to 20.5]
  ALT (SGPT) (U/L)-Day 42 | 14 [12 to 17] | 14 [11 to 19] | 14 [11 to 22] | 13 [10 to 17] | 16 [12 to 25] | 16 [10 to 20] | 15 [11 to 20] | 14 [10 to 19]
  ALT (SGPT) (U/L)-Day 98 | 15 [12 to 17.5] | 15 [12 to 20] | 14.5 [10 to 20] | 14 [10 to 20] | 18 [13 to 26] | 17 [12 to 23] | 15 [12 to 18] | 16 [12 to 23]
  ALT (SGPT) (U/L)-Day 182 | 15 [13 to 18] | 17 [13 to 22] | 14 [11 to 21] | 16 [11 to 20] | 16 [13 to 23.5] | 19.5 [10 to 27] | 16 [11 to 22] | 20 [11 to 27]
  AST (U/L)-Screening | 20 [17 to 22] | 18.5 [16 to 23] | 19 [16 to 23] | 19 [16 to 24] | 20 [17 to 22] | 19 [16 to 24] | 19.5 [16 to 23] | 20 [16.5 to 22.5]
  AST (U/L)-Day 14 | 18 [16.5 to 21] | 18 [15 to 22] | 19 [16 to 25] | 18 [15 to 21] | 19.5 [16 to 23] | 19.5 [15 to 25] | 19 [15 to 22] | 19 [17 to 21.5]
  AST (U/L)-Day 42 | 19.5 [17 to 21] | 19 [16 to 22] | 18 [15 to 22] | 16.5 [14 to 20.5] | 19 [16 to 25] | 19 [15 to 23] | 19 [18 to 22] | 19 [15 to 23]
  AST (U/L)-Day 98 | 17.5 [15.5 to 21] | 18 [16 to 22] | 18.5 [15 to 22] | 18 [15 to 22] | 20 [16 to 23] | 20 [16 to 26] | 18 [15.5 to 22.5] | 20 [18 to 23]
  AST (U/L)-Day 182 | 19 [15.5 to 21.5] | 20 [16 to 24] | 19 [16 to 23] | 18.5 [16 to 26] | 19.5 [17 to 23] | 21 [17 to 27] | 19 [16 to 23] | 23 [18 to 28]
  Alkaline Phosphatase (U/L)-Screening | 60.5 [47 to 71] | 72.5 [60 to 89] | 70.5 [59 to 88] | 70 [54 to 78] | 69.5 [54 to 80] | 70 [55 to 83] | 66 [58 to 85] | 59.5 [55 to 80]
  Alkaline Phosphatase (U/L)-Day 14 | 60.5 [45.5 to 68.5] | 67 [56 to 84] | 62.5 [53 to 89] | 65.5 [49 to 76] | 64 [53 to 80] | 68 [55 to 81.5] | 63 [51 to 77.5] | 65.5 [50.5 to 75.5]
  Alkaline Phosphatase (U/L)-Day 42 | 60 [48 to 68] | 67 [57 to 78] | 67 [55 to 84] | 64 [51.5 to 77.5] | 62 [54 to 81] | 68 [56 to 79] | 65 [51 to 76] | 67 [57 to 80]
  Alkaline Phosphatase (U/L)-Day 98 | 60 [47 to 69] | 64 [60 to 78] | 65 [56 to 84] | 63 [52 to 75] | 62 [52 to 78] | 68 [53 to 77] | 62 [53 to 75] | 66.5 [48 to 82]
  Alkaline Phosphatase (U/L)-Day 182 | 62.5 [50 to 74.5] | 70 [61 to 77] | 70 [57 to 88] | 69 [53 to 85] | 64.5 [52 to 78] | 69.5 [60 to 81] | 65 [57 to 79] | 68 [54 to 85]

12. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine.
Description: as for outcome 11
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 1, 3, and 6
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
mg/dL
  Creatinine (mg/dL)-Screening | 0.795 [0.7 to 0.92] | 0.8 [0.7 to 0.91] | 0.8 [0.7 to 0.89] | 0.79 [0.7 to 0.91] | 0.77 [0.67 to 0.87] | 0.715 [0.62 to 0.87] | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 0.9]
  Creatinine (mg/dL)-Day 14 | 0.785 [0.685 to 0.97] | 0.84 [0.65 to 0.95] | 0.8 [0.7 to 0.87] | 0.88 [0.77 to 0.95] | 0.78 [0.65 to 0.9] | 0.79 [0.7 to 0.88] | 0.8 [0.7 to 0.915] | 0.805 [0.7 to 0.895]
  Creatinine (mg/dL)-Day 42 | 0.83 [0.71 to 0.92] | 0.83 [0.7 to 0.95] | 0.805 [0.7 to 0.9] | 0.81 [0.77 to 0.9] | 0.8 [0.7 to 0.89] | 0.79 [0.63 to 0.9] | 0.8 [0.7 to 0.93] | 0.84 [0.72 to 0.94]
  Creatinine (mg/dL)-Day 98 | 0.815 [0.72 to 0.905] | 0.8 [0.695 to 0.945] | 0.8 [0.7 to 0.94] | 0.81 [0.72 to 0.91] | 0.78 [0.7 to 0.9] | 0.79 [0.7 to 0.81] | 0.83 [0.7 to 0.95] | 0.9 [0.75 to 0.94]
  Creatinine (mg/dL)-Day 182 | 0.81 [0.7 to 0.93] | 0.855 [0.72 to 0.98] | 0.8 [0.7 to 0.93] | 0.84 [0.76 to 0.98] | 0.8 [0.7 to 0.9] | 0.785 [0.7 to 0.9] | 0.84 [0.7 to 1] | 0.87 [0.8 to 0.93]

13. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin.
Description: as for outcome 11
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 1, 3, and 6
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
g/dL
  Hemoglobin (g/dL)-Screening | 14.15 [12.6 to 14.9] | 14.3 [13.3 to 15.5] | 14.2 [13 to 15.4] | 14.2 [13.5 to 15.5] | 14.2 [13.5 to 15.3] | 14.5 [12.9 to 15.3] | 13.85 [13.3 to 15.3] | 14.6 [12.95 to 15.15]
  Hemoglobin (g/dL)-Day 14 | 13.6 [12.6 to 14.4] | 13.8 [13.2 to 14.8] | 13.6 [12.4 to 14.7] | 13.55 [12.6 to 15] | 13.9 [12.7 to 14.9] | 13.7 [12.1 to 14.65] | 13.4 [12.85 to 14.5] | 14.05 [12.5 to 14.5]
  Hemoglobin (g/dL)-Day 42 | 13.6 [13 to 15.1] | 13.8 [12.9 to 14.8] | 13.8 [12.7 to 14.8] | 13.75 [12.75 to 14.7] | 13.9 [13.3 to 15.2] | 14 [12.5 to 15] | 13.9 [13 to 14.5] | 14 [13.1 to 14.7]
  Hemoglobin (g/dL)-Day 98 | 13.5 [12.8 to 15.2] | 13.95 [12.75 to 15.25] | 13.9 [13.1 to 15] | 13.7 [12.9 to 15.1] | 14.1 [13.1 to 15.4] | 14.05 [12.8 to 15] | 14 [13.2 to 15] | 14.35 [12.6 to 14.9]
  Hemoglobin (g/dL)-Day 182 | 13.75 [13.2 to 15.05] | 14 [13.4 to 15.3] | 14.1 [13.2 to 15.4] | 14 [12.9 to 15.2] | 14.03 [12.6 to 15] | 14.05 [13 to 15] | 14.05 [13.5 to 15] | 14.1 [13.4 to 15.2]

14. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocytes, Neutrophils.
Description: as for outcome 11
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 1, 3, and 6
Measure: Median (Inter-Quartile Range); unit: cells/cubic mm
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
cells/cubic mm
  Neutrophils (cells/cubic mm)-Screening | 4060.5 [2740 to 5069] | 3540 [2870 to 4352] | 3108.5 [2670 to 4498] | 3919 [3280 to 4627] | 3616 [2725 to 4718] | 3505 [2719 to 4269] | 3389 [2684 to 4397] | 3861 [2953.5 to 4597.5]
  Neutrophils (cells/cubic mm)-Day 14 | 3156.5 [2499 to 4400.5] | 3230 [2437 to 3830] | 3404 [2353 to 4158] | 3108 [2717 to 4623] | 3910 [2614 to 4854] | 3874 [2840.5 to 5127.5] | 3420 [2535 to 4515.5] | 3366.5 [2682 to 5314]
  Neutrophils (cells/cubic mm)-Day 42 | 3149 [2840 to 4349] | 2795 [2255.5 to 4220] | 3300 [2448 to 4250] | 3467.5 [2790 to 4144] | 3440 [2773 to 4370] | 3580 [2740 to 4370] | 3630 [2805 to 4678] | 3532 [2729 to 4910]
  Neutrophils (cells/cubic mm)-Day 98 | 2980 [2310 to 4002] | 2969 [2272 to 3763.5] | 3602.5 [2622 to 4310] | 3805 [3103 to 4540] | 3519 [2904 to 4193] | 3331.5 [2730 to 4482] | 3345 [2542 to 3928] | 3433 [2656 to 4110]
  Neutrophils (cells/cubic mm)-Day 182 | 3061 [2815.5 to 4376.5] | 3259 [2562 to 4132] | 3311 [2636 to 4534] | 3508.5 [2754 to 4863] | 3616 [2840 to 4863] | 3395 [2758 to 4190] | 3794.5 [2897 to 5210] | 3370 [2738 to 3926]
  Lymphocytes (cells/cubic mm)-Screening | 2033 [1660 to 2590] | 1906 [1670 to 2470] | 2044.5 [1730 to 2405] | 1993.5 [1610 to 2310] | 2054.5 [1550 to 2412] | 2002.5 [1740 to 2384] | 1942 [1570 to 2270] | 2150 [1940.5 to 2796.5]
  Lymphocytes (cells/cubic mm)-Day 14 | 1963.5 [1578 to 2269.5] | 1953 [1587 to 2469] | 1936 [1593 to 2283] | 1965 [1699 to 2440] | 1857 [1600 to 2356] | 2014.5 [1621 to 2303] | 1746.5 [1540 to 2138] | 2030.5 [1891 to 2296.5]
  Lymphocytes (cells/cubic mm)-Day 42 | 1881.5 [1611 to 2150] | 1794 [1430 to 2488] | 1972 [1681 to 2320] | 1944 [1720 to 2465] | 2060 [1784 to 2640] | 1990 [1752 to 2267] | 1910 [1556 to 2400] | 2008 [1650 to 2450]
  Lymphocytes (cells/cubic mm)-Day 98 | 1859 [1570 to 2111] | 1920.5 [1599.5 to 2135.5] | 2010 [1722 to 2332] | 2035 [1651 to 2550] | 2003 [1660 to 2330] | 1907.5 [1653 to 2180] | 1863 [1640 to 2230] | 2198 [1922 to 2613]
  Lymphocytes (cells/cubic mm)-Day 182 | 1868 [1385 to 2175] | 1887 [1590 to 2309] | 1848.5 [1550 to 2264] | 2090.5 [1566 to 2400] | 1990 [1810 to 2570] | 2066.5 [1683 to 2310] | 1795 [1522 to 2291] | 1962 [1806.5 to 2569]

15. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC.
Description: as for outcome 11
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 1, 3, and 6
Measure: Median (Inter-Quartile Range); unit: x1000/cubic mm
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
x1000/cubic mm
  WBC (x1000/cubic mm)-Screening | 6.53 [5.57 to 8.27] | 6.45 [5.3 to 7.32] | 5.94 [4.92 to 7.87] | 6.665 [5.72 to 7.2] | 6.35 [5.17 to 7.6] | 5.94 [5.17 to 7.66] | 6.17 [5.3 to 6.81] | 7.135 [5.705 to 8.08]
  WBC (x1000/cubic mm)-Day 14 | 5.705 [5.06 to 6.905] | 6.04 [4.68 to 7.1] | 5.795 [4.64 to 6.86] | 6.155 [5.05 to 6.9] | 6.41 [4.96 to 7.85] | 6.25 [5.25 to 8.225] | 6 [5.11 to 7.17] | 6.36 [5.37 to 7.96]
  WBC (x1000/cubic mm)-Day 42 | 5.815 [5 to 7.24] | 5.55 [4.6 to 7.1] | 6 [4.68 to 7.2] | 6.04 [5.265 to 7.4] | 6.25 [5.3 to 7.63] | 6.4 [5.34 to 7.26] | 6.09 [5.38 to 7.4] | 6.9 [5.2 to 8]
  WBC (x1000/cubic mm)-Day 98 | 5.92 [4.56 to 6.4] | 5.69 [4.635 to 6.705] | 5.985 [5.02 to 7.34] | 6.68 [5.91 to 7.48] | 6.22 [5.02 to 7.3] | 6.075 [5.28 to 7.24] | 5.8 [5.2 to 6.9] | 6.41 [5.4 to 6.92]
  WBC (x1000/cubic mm)-Day 182 | 5.6 [4.875 to 7.345] | 6.29 [5 to 7.4] | 5.515 [5.1 to 7.36] | 6.46 [5.31 to 7.6] | 6.39 [5.44 to 7.6] | 5.9 [5.31 to 7.35] | 6.585 [5.5 to 7.54] | 5.835 [5.31 to 7.42]
  Platelets (x1000/cubic mm)-Screening | 232.5 [199 to 311] | 243 [216 to 296] | 269.5 [226 to 304] | 258 [228 to 291] | 275 [225 to 314] | 280 [240 to 303] | 264.5 [238 to 288] | 252.5 [226.5 to 303]
  Platelets (x1000/cubic mm)-Day 14 | 223.5 [201.5 to 281.5] | 236 [215 to 299] | 264.5 [218.4 to 311] | 255.15 [233 to 291] | 285 [245 to 318] | 279.5 [249 to 318.5] | 284 [249 to 310.5] | 257.5 [230 to 289.5]
  Platelets (x1000/cubic mm)-Day 42 | 222.5 [206.6 to 282] | 241 [210 to 285] | 264 [204 to 303] | 258.95 [242 to 310.85] | 292 [250 to 331] | 288 [247 to 320] | 286 [251 to 334] | 248 [227.5 to 299]
  Platelets (x1000/cubic mm)-Day 98 | 241 [200.9 to 287] | 250.5 [213.2 to 318] | 271 [220 to 334] | 254 [224 to 289] | 258 [228 to 291] | 259 [230 to 290] | 260 [232 to 292] | 262.75 [218 to 284.8]
  Platelets (x1000/cubic mm)-Day 182 | 238.5 [198.5 to 276] | 265.9 [224 to 309] | 269.5 [230 to 324] | 256.2 [232 to 288] | 284 [240 to 327] | 276 [244 to 306] | 279 [246 to 315] | 257.5 [237.5 to 293]

16. Primary Outcome: Numbers of Participants With Grade 1 or Higher Local Laboratory Results.
Description: The numbers (percentages) of participants with local laboratory values recorded as meeting Grade 1 AE criteria or above as specified in the DAIDS AE Grading Table were tabulated by treatment group for each post vaccination timepoint.
Time Frame: Measured during screening, and 2 weeks after each vaccination at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 30 | 50 | 50 | 30 | 50 | 50 | 50 | 24
Participants
  Lymphocytes (cells/cubic mm)-Day 98 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets (x1000/cubic mm)-Day 14 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)-Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine (mg/dL)-Day 14 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Creatinine (mg/dL)-Day 42 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Creatinine (mg/dL)-Day 98 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1
  Creatinine (mg/dL)-Day 182 | 0 | 4 | 1 | 2 | 3 | 1 | 2 | 1

17. Primary Outcome: Occurrence and Level of HIV-specific Total IgG Binding Antibody Response Breadth and Magnitude - Positive Response Rates.
Description: IgG binding antibody breadth assays were not run. Instead, IgG was assayed against a smaller panel of antigens. Serum IgG responses were measured on a Bio-Plex instrument using a custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen minus reference antigen MFI. Net MFI below 1 is set to 1, and Net MFI above 22,000 is set to 22,000. Samples from post-baseline visits have positive responses if they meet three criteria: (1) net MFI >= antigen-specific threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI > 3 times baseline net MFI, and (3) experimental antigen MFI > 3 times baseline MFI. Data are excluded if the blood draw date was outside the allowable window, a participant was HIV-infected, or the reference antigen exceeds 5000 MFI.
Time Frame: Measured at Month 6.5
Population: In this report, the "overall number of participants analyzed" represents the HIV uninfected participants with specimens at Month6.5. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available BAMA data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
Participants
  00MSA 4076 gp140: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  00MSA 4076 gp140 | 19 | 41 | 42 | 24 | 39 | 33 | 38 | 0
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  1086C_D7gp120.avi/293F | 19 | 44 | 44 | 24 | 39 | 35 | 39 | 1
  96ZM651.gp140C.avi: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  96ZM651.gp140C.avi | 19 | 42 | 42 | 24 | 39 | 34 | 38 | 0
  A1.con.env03 140 CF: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  A1.con.env03 140 CF | 19 | 41 | 42 | 24 | 39 | 34 | 37 | 0
  Con 6 gp120/B: number analyzed (Participants) | 21 | 44 | 44 | 25 | 39 | 35 | 40 | 18
  Con 6 gp120/B | 19 | 41 | 42 | 24 | 36 | 33 | 36 | 0
  Con S gp140 CFI: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  Con S gp140 CFI | 20 | 42 | 42 | 24 | 39 | 35 | 39 | 0

18. Primary Outcome: Occurrence and Level of HIV-specific Total IgG Binding Antibody Response Breadth and Magnitude - Magnitudes.
Description: IgG binding antibody breadth assays were not run. Instead, IgG was assayed against a smaller panel of antigens.Serum IgG responses were measured on a Bio-Plex instrument using a custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen minus reference antigen MFI. Net MFI below 1 is set to 1, and Net MFI above 22,000 is set to 22,000. Samples from post-baseline visits have positive responses if they meet three criteria: (1) net MFI >= antigen-specific threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI > 3 times baseline net MFI, and (3) experimental antigen MFI > 3 times baseline MFI. Data are excluded if the blood draw date was outside the allowable window, a participant was HIV-infected, or the reference antigen exceeds 5000 MFI.
Time Frame: Measured at Month 6.5
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
relative fluorescence units
  00MSA 4076 gp140: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  00MSA 4076 gp140 | 22000 [11213.5 to 22000] | 22000 [22000 to 22000] | 22000 [15544.625 to 22000] | 22000 [14452.5 to 22000] | 22000 [22000 to 22000] | 22000 [21484.5 to 22000] | 22000 [22000 to 22000] | 1 [1 to 1]
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  1086C_D7gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1 [1 to 5]
  96ZM651.gp140C.avi: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  96ZM651.gp140C.avi | 21251 [11922.5 to 22000] | 22000 [22000 to 22000] | 22000 [21760.75 to 22000] | 22000 [17409.5 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1 [1 to 1]
  A1.con.env03 140 CF: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  A1.con.env03 140 CF | 22000 [15131.25 to 22000] | 22000 [20624.625 to 22000] | 22000 [15995.5 to 22000] | 22000 [13013 to 22000] | 22000 [22000 to 22000] | 22000 [19209.125 to 22000] | 22000 [22000 to 22000] | 1 [1 to 1]
  Con 6 gp120/B: number analyzed (Participants) | 21 | 44 | 44 | 25 | 39 | 35 | 40 | 18
  Con 6 gp120/B | 22000 [10550 to 22000] | 22000 [22000 to 22000] | 22000 [18086.25 to 22000] | 22000 [16341.75 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [20235.75 to 22000] | 9.75 [1 to 62]
  Con S gp140 CFI: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  Con S gp140 CFI | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1 [1 to 4.25]

19. Primary Outcome: Occurrence and Level of Anti -V1/V2 Scaffold IgG Binding Antibody Responses - Positive Response Rates.
Description: Serum IgG responses were measured on a Bio-Plex instrument using a custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen minus reference antigen MFI. Net MFI below 1 is set to 1, and Net MFI above 22,000 is set to 22,000. Samples from post-baseline visits have positive responses if they meet three criteria: (1) net MFI >= antigen-specific threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI > 3 times baseline net MFI, and (3) experimental antigen MFI > 3 times baseline MFI. Data are excluded if the blood draw date was outside the allowable window, a participant was HIV-infected, or the reference antigen exceeds 5000 MFI.
Time Frame: Measured at Month 6.5
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
Participants
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  TV1c8_D11gp120.avi/293F | 19 | 42 | 43 | 24 | 39 | 36 | 40 | 0
  gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 21 | 44 | 44 | 25 | 39 | 34 | 40 | 17
  gp70-TV1.GSKvacV1V2/293F | 16 | 35 | 24 | 23 | 35 | 31 | 30 | 0
  gp70_B.CaseA_V1_V2: number analyzed (Participants) | 21 | 44 | 43 | 25 | 38 | 34 | 40 | 17
  gp70_B.CaseA_V1_V2 | 16 | 31 | 20 | 22 | 33 | 30 | 28 | 0

20. Primary Outcome: Occurrence and Level of Anti -V1/V2 Scaffold IgG Binding Antibody Response - Magnitudes.
Description: as for outcome 19
Time Frame: Measured at Month 6.5
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
relative fluorescence units
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 21 | 44 | 44 | 25 | 40 | 36 | 40 | 18
  TV1c8_D11gp120.avi/293F | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1 [1 to 26.75]
  gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 21 | 44 | 44 | 25 | 39 | 34 | 40 | 17
  gp70-TV1.GSKvacV1V2/293F | 521.5 [113.75 to 6977.75] | 1656 [136 to 11641.600001] | 330 [1 to 1337.25] | 4948.75 [1574.25 to 11707.75] | 16511.5 [2093 to 22000] | 10392.25 [1706.5 to 22000] | 2409 [317.125 to 16400.5] | 1 [1 to 1]
  gp70_B.CaseA_V1_V2: number analyzed (Participants) | 21 | 44 | 43 | 25 | 38 | 34 | 40 | 17
  gp70_B.CaseA_V1_V2 | 744.5 [148.75 to 7460.75] | 1110.625 [86.125 to 7316.5] | 184.5 [1 to 1269.75] | 1881 [589 to 6311] | 5559 [1255 to 18096.5] | 5231.875 [1003.5 to 10415.25] | 1329.625 [179.625 to 8718] | 1 [1 to 1]

21. Primary Outcome: Occurrence and Level of Neutralizing Antibody Responses Against HIV-1 Isolates.
Description: The neutralizing antibody assay was not run. Therefore this dataset doesn't exist
Time Frame: Measured at Month 6.5
Population: Data were not collected
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Primary Outcome: Occurrence and Level of HIV-specific CD4+ T-cell Responses - Positive Response Rates.
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if p<=0.00001. Any Env magnitude is the maximum of gp120 and Env ZM96 magnitude; Any Pol is the sum of CN54 magnitude; and Any HIV is the sum of Gag ZM96, Nef CN54, Any Pol, and Any Env. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high.
Time Frame: Measured at Month 6.5
Population: In this report, the "overall number of participants analyzed" represents the HIV uninfected participants with specimens at Month6.5. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available ICS data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
Participants
  ANY HIV: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  ANY HIV | 20 | 47 | 43 | 21 | 42 | 40 | 40 | 1
  ANY ENV: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  ANY ENV | 20 | 47 | 42 | 20 | 42 | 40 | 40 | 1
  ANY POL: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  ANY POL | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 1
  Env-1-ZM96: number analyzed (Participants) | 23 | 48 | 43 | 25 | 43 | 40 | 41 | 20
  Env-1-ZM96 | 16 | 41 | 40 | 12 | 32 | 34 | 26 | 1
  Env-2-ZM96: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  Env-2-ZM96 | 12 | 25 | 28 | 5 | 18 | 21 | 16 | 1
  Gag-ZM96: number analyzed (Participants) | 23 | 48 | 43 | 25 | 43 | 40 | 42 | 20
  Gag-ZM96 | 9 | 14 | 10 | 3 | 5 | 8 | 4 | 1
  Nef-CN54: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  Nef-CN54 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Pol-1-CN54: number analyzed (Participants) | 23 | 48 | 43 | 26 | 42 | 40 | 42 | 20
  Pol-1-CN54 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Pol-2-CN54: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  Pol-2-CN54 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
  TV1 gp120: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  TV1 gp120 | 17 | 47 | 42 | 17 | 41 | 39 | 38 | 1
  1086 gp120: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  1086 gp120 | 17 | 47 | 42 | 17 | 38 | 40 | 39 | 1

23. Primary Outcome: Occurrence and Level of HIV-specific CD4+ T-cell Responses - Magnitudes.
Description: as for outcome 22
Time Frame: Measured at Month 6.5
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: percent T-cells
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
percent T-cells
  ANY HIV: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  ANY HIV | 0.237 [0.084 to 0.437] | 0.388 [0.245 to 0.521] | 0.492 [0.334 to 0.827] | 0.156 [0.06 to 0.253] | 0.364 [0.187 to 0.495] | 0.48 [0.334 to 0.681] | 0.52 [0.209 to 0.69] | 0.016 [-0.013 to 0.036]
  ANY ENV: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  ANY ENV | 0.189 [0.076 to 0.332] | 0.37 [0.228 to 0.485] | 0.451 [0.334 to 0.829] | 0.124 [0.054 to 0.227] | 0.328 [0.167 to 0.484] | 0.456 [0.357 to 0.65] | 0.504 [0.202 to 0.741] | 0.015 [0.006 to 0.02]
  ANY POL: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  ANY POL | 0.003 [-0.009 to 0.01] | -0.001 [-0.011 to 0.007] | 0 [-0.016 to 0.01] | 0.003 [-0.008 to 0.01] | -0.001 [-0.009 to 0.011] | -0.002 [-0.017 to 0.01] | -0.002 [-0.01 to 0.005] | 0.001 [-0.009 to 0.01]
  Env-1-ZM96: number analyzed (Participants) | 23 | 48 | 43 | 25 | 43 | 40 | 41 | 20
  Env-1-ZM96 | 0.076 [0.038 to 0.21] | 0.196 [0.117 to 0.305] | 0.272 [0.14 to 0.445] | 0.038 [0.021 to 0.072] | 0.12 [0.054 to 0.155] | 0.186 [0.092 to 0.261] | 0.092 [0.033 to 0.232] | 0.008 [-0.001 to 0.015]
  Env-2-ZM96: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  Env-2-ZM96 | 0.047 [0.016 to 0.104] | 0.052 [0.031 to 0.088] | 0.085 [0.038 to 0.161] | 0.02 [0.009 to 0.025] | 0.04 [0.015 to 0.108] | 0.054 [0.019 to 0.095] | 0.045 [0.015 to 0.097] | 0 [-0.004 to 0.008]
  Gag-ZM96: number analyzed (Participants) | 23 | 48 | 43 | 25 | 43 | 40 | 42 | 20
  Gag-ZM96 | 0.039 [0.013 to 0.066] | 0.027 [0.014 to 0.05] | 0.03 [0.013 to 0.054] | 0.016 [0.011 to 0.022] | 0.011 [0.001 to 0.025] | 0.013 [0.006 to 0.045] | -0.002 [-0.009 to 0.009] | 0.001 [-0.006 to 0.006]
  Nef-CN54: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  Nef-CN54 | -0.003 [-0.005 to 0.003] | -0.001 [-0.008 to 0.003] | -0.002 [-0.014 to 0.004] | 0 [-0.006 to 0.003] | -0.004 [-0.01 to 0.001] | -0.004 [-0.012 to 0.004] | -0.001 [-0.009 to 0.007] | -0.002 [-0.008 to 0.002]
  Pol-1-CN54: number analyzed (Participants) | 23 | 48 | 43 | 26 | 42 | 40 | 42 | 20
  Pol-1-CN54 | 0.001 [-0.005 to 0.004] | -0.001 [-0.007 to 0.004] | 0 [-0.007 to 0.005] | 0.001 [-0.004 to 0.008] | 0.001 [-0.006 to 0.005] | 0 [-0.007 to 0.004] | -0.001 [-0.006 to 0.003] | -0.001 [-0.005 to 0.002]
  Pol-2-CN54: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  Pol-2-CN54 | -0.001 [-0.006 to 0.008] | -0.002 [-0.008 to 0.005] | -0.001 [-0.012 to 0.009] | 0.001 [-0.004 to 0.006] | -0.002 [-0.009 to 0.006] | -0.003 [-0.008 to 0.006] | -0.001 [-0.005 to 0.006] | 0.001 [-0.005 to 0.008]
  TV1 gp120: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  TV1 gp120 | 0.151 [0.049 to 0.309] | 0.349 [0.193 to 0.47] | 0.319 [0.215 to 0.625] | 0.096 [0.041 to 0.227] | 0.271 [0.152 to 0.421] | 0.376 [0.284 to 0.504] | 0.334 [0.201 to 0.578] | -0.003 [-0.008 to -0.002]
  1086 gp120: number analyzed (Participants) | 23 | 48 | 43 | 26 | 43 | 40 | 42 | 20
  1086 gp120 | 0.123 [0.037 to 0.278] | 0.308 [0.159 to 0.373] | 0.448 [0.272 to 0.751] | 0.078 [0.029 to 0.135] | 0.241 [0.116 to 0.393] | 0.412 [0.273 to 0.566] | 0.42 [0.132 to 0.651] | -0.001 [-0.006 to 0.007]

24. Primary Outcome: Occurrence and Level of HIV-specific CD8+ T-cell Responses - Positive Response Rates.
Description: as for outcome 22
Time Frame: Measured at Month 6.5
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
Participants
  ANY HIV: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  ANY HIV | 2 | 2 | 11 | 1 | 4 | 6 | 4 | 1
  ANY ENV: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  ANY ENV | 2 | 1 | 9 | 1 | 2 | 5 | 4 | 1
  ANY POL: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  ANY POL | 0 | 0 | 3 | 0 | 2 | 1 | 1 | 1
  Env-1-ZM96: number analyzed (Participants) | 23 | 49 | 44 | 25 | 43 | 40 | 41 | 19
  Env-1-ZM96 | 1 | 1 | 3 | 1 | 0 | 3 | 2 | 1
  Env-2-ZM96: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Env-2-ZM96 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0
  Gag-ZM96: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Gag-ZM96 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0
  Nef-CN54: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Nef-CN54 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pol-1-CN54: number analyzed (Participants) | 23 | 49 | 44 | 26 | 42 | 40 | 42 | 19
  Pol-1-CN54 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  Pol-2-CN54: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Pol-2-CN54 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
  TV1 gp120: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  TV1 gp120 | 1 | 0 | 2 | 0 | 1 | 4 | 2 | 1
  1086 gp120: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  1086 gp120 | 1 | 0 | 2 | 0 | 0 | 2 | 2 | 1

25. Primary Outcome: Occurrence and Level of HIV-specific CD8+ T-cell Responses - Magnitudes.
Description: as for outcome 22
Time Frame: Measured at Month 6.5
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: percent T-cells
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
Number analyzed (Participants) | 23 | 49 | 46 | 26 | 43 | 42 | 42 | 21
percent T-cells
  ANY HIV: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  ANY HIV | 0.007 [-0.004 to 0.035] | 0.019 [-0.001 to 0.042] | 0.026 [0.007 to 0.062] | 0.012 [-0.004 to 0.021] | 0.019 [0.001 to 0.043] | 0.006 [-0.002 to 0.044] | 0.013 [0.002 to 0.044] | -0.004 [-0.011 to 0.009]
  ANY ENV: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  ANY ENV | 0.006 [-0.001 to 0.014] | 0.011 [0.003 to 0.019] | 0.013 [0.004 to 0.037] | 0.01 [0.003 to 0.021] | 0.008 [0.002 to 0.032] | 0.009 [0.005 to 0.022] | 0.009 [0.003 to 0.02] | 0.004 [-0.001 to 0.009]
  ANY POL: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  ANY POL | -0.002 [-0.006 to 0.001] | 0.002 [-0.005 to 0.013] | 0.002 [-0.006 to 0.01] | -0.001 [-0.007 to 0.003] | -0.001 [-0.005 to 0.005] | 0 [-0.009 to 0.006] | 0 [-0.004 to 0.007] | -0.005 [-0.011 to 0.002]
  Env-1-ZM96: number analyzed (Participants) | 23 | 49 | 44 | 25 | 43 | 40 | 41 | 19
  Env-1-ZM96 | -0.001 [-0.005 to 0.002] | 0.003 [-0.003 to 0.01] | 0.002 [-0.003 to 0.01] | 0.001 [-0.005 to 0.005] | 0.005 [-0.002 to 0.014] | 0.005 [0 to 0.015] | 0.006 [0.002 to 0.012] | -0.003 [-0.006 to 0.005]
  Env-2-ZM96: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Env-2-ZM96 | 0.001 [-0.002 to 0.005] | 0.002 [-0.003 to 0.007] | 0 [-0.003 to 0.007] | 0.005 [0 to 0.01] | 0 [-0.003 to 0.007] | -0.002 [-0.004 to 0.008] | 0 [-0.004 to 0.006] | -0.002 [-0.005 to 0.001]
  Gag-ZM96: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Gag-ZM96 | 0.002 [-0.002 to 0.007] | 0.001 [-0.003 to 0.006] | 0.003 [0 to 0.011] | 0 [-0.003 to 0.004] | 0.002 [-0.002 to 0.006] | 0.001 [-0.002 to 0.01] | 0.002 [-0.003 to 0.007] | -0.001 [-0.004 to 0]
  Nef-CN54: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Nef-CN54 | -0.003 [-0.004 to 0] | 0 [-0.004 to 0.005] | 0.001 [-0.005 to 0.005] | 0 [-0.003 to 0.003] | -0.001 [-0.005 to 0.004] | -0.002 [-0.005 to 0.001] | -0.001 [-0.004 to 0.006] | -0.003 [-0.006 to 0.002]
  Pol-1-CN54: number analyzed (Participants) | 23 | 49 | 44 | 26 | 42 | 40 | 42 | 19
  Pol-1-CN54 | -0.003 [-0.004 to 0] | 0.001 [-0.003 to 0.003] | 0.002 [-0.004 to 0.006] | -0.002 [-0.004 to 0.002] | 0 [-0.003 to 0.002] | 0 [-0.004 to 0.004] | 0.001 [-0.002 to 0.004] | 0 [-0.005 to 0.003]
  Pol-2-CN54: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  Pol-2-CN54 | 0 [-0.003 to 0.001] | 0.001 [-0.002 to 0.004] | 0.001 [-0.003 to 0.005] | 0 [-0.005 to 0.004] | -0.001 [-0.005 to 0.003] | 0 [-0.007 to 0.003] | 0 [-0.003 to 0.005] | -0.003 [-0.005 to 0]
  TV1 gp120: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  TV1 gp120 | 0 [-0.005 to 0.004] | 0.002 [-0.004 to 0.007] | 0.002 [-0.005 to 0.008] | 0.001 [-0.004 to 0.006] | 0.003 [-0.003 to 0.012] | 0.003 [-0.003 to 0.009] | 0.001 [-0.002 to 0.004] | 0 [-0.005 to 0.005]
  1086 gp120: number analyzed (Participants) | 23 | 49 | 44 | 26 | 43 | 40 | 42 | 19
  1086 gp120 | 0.003 [-0.002 to 0.01] | 0.002 [-0.003 to 0.01] | 0.002 [-0.004 to 0.014] | 0.005 [-0.002 to 0.013] | 0.001 [-0.003 to 0.014] | 0.001 [-0.003 to 0.009] | 0 [-0.004 to 0.009] | -0.001 [-0.006 to 0.004]

ADVERSE EVENTS:
Time Frame: Serious adverse events and new chronic conditions requiring medical intervention of more than 30 days were collected through the month 12 timepoint. Adverse events of special interest were collected through month 18. All other AEs were collected through 30 days after each vaccination.
Description: Adverse events of special interest were described in the protocol Appendix J. AESI for this protocol include but are not limited to potential immune-mediated diseases.
Arm/Group | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B | Group 7: Placebo + Protein/AS01B | Group 8: Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/50 | 0/50 | 0/30 | 0/50 | 0/50 | 0/50 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/50 | 0/50 | 1/30 | 1/50 | 1/50 | 0/50 | 0/24
Other Adverse Events (participants affected / at risk) | 24/30 | 33/50 | 34/50 | 20/30 | 39/50 | 31/50 | 27/50 | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 (N=30) | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 (N=30) | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 7: Placebo + Protein/AS01B (N=50) | Group 8: Placebo (N=24)
Any SOC (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DNA-HIV-PT123 + Placebo + Protein/MF59 (N=30) | Group 2: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 3: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 4: DNA-HIV-PT123 + Placebo + Protein/MF59 (N=30) | Group 5: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 6: DNA-HIV-PT123 + Placebo + Protein/AS01B (N=50) | Group 7: Placebo + Protein/AS01B (N=50) | Group 8: Placebo (N=24)
Any SOC (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Any SOC (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Gastrointestinal disorders) | 2 (7) | 4 (4) | 4 (4) | 1 (1) | 2 (4) | 5 (5) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any SOC (General disorders) | 1 (1) | 4 (4) | 4 (4) | 4 (5) | 5 (7) | 1 (1) | 3 (3) | 1 (1)
Axillary pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hangover (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any SOC (Infections and infestations) | 12 (14) | 15 (19) | 20 (32) | 7 (10) | 21 (24) | 16 (23) | 12 (15) | 8 (10)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (4) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Genitourinary tract gonococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycetoma mycotic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 8 (8) | 8 (8) | 3 (3) | 13 (13) | 8 (8) | 7 (7) | 6 (6)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginitis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Viral rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 5 (5) | 1 (2) | 4 (4) | 1 (1) | 4 (4) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Investigations) | 1 (1) | 10 (17) | 8 (11) | 5 (6) | 15 (22) | 8 (16) | 5 (9) | 5 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 7 (11) | 3 (6) | 2 (2) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 4 (5) | 3 (3) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 6 (6) | 4 (5) | 3 (3) | 4 (4) | 2 (5) | 3 (4) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2) | 4 (4) | 3 (3) | 4 (9) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Any SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Nervous system disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 3 (4) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (2) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Any SOC (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any SOC (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Alcoholic hangover (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Any SOC (Renal and urinary disorders) | 2 (3) | 4 (7) | 2 (2) | 3 (4) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Any SOC (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Any SOC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any SOC (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (4) | 3 (4) | 3 (3) | 6 (6) | 6 (8) | 3 (3) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any SOC (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT02915016/Prot_SAP_ICF_000.pdf